CLINICAL TRIAL: NCT04692805
Title: EUS-guided Partial Splenic Embolization in Combination With EUS-guided Treatment of Varices for Patients With Portal Hypertension
Brief Title: EUS-guided PSE in Combination With EUS-guided Treatment of Varices for Patients With Portal Hypertension
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tongji Hospital (Other)
Responsible Party: Principal Investigator, Qian Chen, Professor, Tongji Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: S320
Record Dates: First submitted 2020-12-29; First posted 2021-01-05 (Actual); Last update posted 2021-01-08 (Actual); Status verified 2021-01

CONDITIONS: Gastroesophageal Varices; Hypersplenism; Portal Hypertension
MeSH Terms: conditions — Hypersplenism; Hypertension, Portal | interventions — MK 6 cyanoacrylate

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EUS-guided treatment of varices (Experimental): Procedure: EUS-guided injection of coils with cyanoacrylate glue (CYA) and sclerosing agent.
  First CT scan will be ordered to determine the patient having esophageal and gastric varices and splenomegaly.
  Complete blood count (CBC) will be ordered to confirm the deficiency of one or more blood cell lines.
  A standard diagnostic upper endoscopy will be performed in order to classify the varices according to the classification of Sarin and Kumar. Only GOV II and IGV I varices will be included. Once the patient considered as a candidate will be treated with Coils plus CYA and sclerosing agent (Group A).
  Interventions: Device: coils; Drug: cyanoacrylate glue
- EUS-guided partial splenic embolization + EUS-guided treatment of varices (Experimental): Procedure: EUS-guided partial splenic embolization + EUS-guided treatment of varices First CT scan will be ordered to determine the patient having esophageal and gastric varices and splenomegaly.
  Complete blood count (CBC) will be ordered to confirm the deficiency of one or more blood cell lines.
  A standard diagnostic upper endoscopy will be performed in order to classify the varices according to the classification of Sarin and Kumar. Only GOV II and IGV I varices will be included. Once the patient considered as a candidate will be treated with coils plus CYA and sclerosing agent.
  At the same procedure, a branch of splenic artery will be identified by EUS and implanted with coils plus CYA (Group B).
  Interventions: Device: coils; Drug: cyanoacrylate glue

INTERVENTIONS:
Device: coils — EUS-guided injection of coils
Drug: cyanoacrylate glue — EUS-guided injection of cyanoacrylate glue

SUMMARY:
This study aims to evaluate the efficiency of EUS-guided combination therapy (EUS-guided PSE + EUS-guided treatment of varices) to EUS-guided treatment of varices alone in cirrhotic patients with portal hypertension who have developed gastroesophageal variceal hemorrhage and accompanied with hypersplenism.

DETAILED DESCRIPTION:
Partial splenic embolization (PSE) was developed in the purpose of managing two common complications of portal hypertension including variceal bleeding and hypersplenism. The procedure is normally performed by clinicians engaged in interventional radiology via a transcatheter embolization method as the successful embolization of the selected splenic arteries results in devascularization of a focal lesion followed by splenic infarction and subsequently reducing the splenic contribution to the portal blood flow. Our previous case study suggests implanting coil in a branch of splenic artery under the endoscopic ultrasound (EUS) -guidance followed by the glue injection was an alternative PSE procedure to control hypersplenism. Recent advance has also heightened the therapeutic aspect of EUS in managing varices. We have established the novel approach to manage varices and hypersplenism at the same time by combining EUS-guided PSE and EUS-guided treatment of varices. This study aims to evaluate the efficiency of EUS-guided combination therapy (EUS-guided PSE + EUS-guided treatment of varices) to EUS-guided treatment of varices alone in cirrhotic patients with portal hypertension who have developed gastroesophageal variceal hemorrhage and accompanied with hypersplenism.

ELIGIBILITY:
Inclusion Criteria:

* At the risk of gastroesophageal variceal hemorrhage; Acute gastroesophageal variceal hemorrhage; Hematemesis and/or melena resulted from gastroesophageal variceal hemorrhage of liver cirrhosis in the past.
* Hypersplenism is indicated by either abdominal ultrasound or CT image showing splenic enlargement or splenomegaly and CBC test showing deficiency of one or more blood cell lines.
* Consent form must be signed by patients or their guardians before entering the test.

Exclusion Criteria:

* History of liver surgery or spleen surgery and liver cancer
* Coagulopathy (INR > 1.5) or having been taken oral anticoagulation agents such as aspirin, warfarin, etc. in the past week.
* Existence of gastrointestinal endoscopic therapy contraindication; Hemorrhagic shock has not be corrected; Hepatic encephalopathy; Moderate to severe ascites, Poor liver function (Child - Pugh class C).
* Severe cardiorespiratory dysfunction, including sinus bradycardia, bronchial asthma, chronic obstructive pulmonary disease, heart failure, and atrioventricular block
* Pregnant women and nursing mothers.
* Absence of informed consent

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2021-01-05 (Actual); Primary Completion 2021-07-05 (Estimated); Study Completion 2022-01-05 (Estimated)

PRIMARY OUTCOMES:
Efficacy of EUS-guided treatment for varices | 6 months
  Efficacy will be determined by recording recurrent events of hematemesis and/or melena after the EUS-guided procedure. Further confirmation of gastroesophageal variceal hemorrhage will be evaluated by upper gastric endoscopy and lab tests.

SECONDARY OUTCOMES:
Safety of EUS-guided combination therapy in cirrhotic patients with gastroesophageal varices and hypersplenism | 6 months
  Safety will be determined by measure of incidence of adverse events related to EUS-guided procedure within and after 30 days of the procedure.
Efficacy of EUS-guided partial splenic embolization | 6 months
  Efficacy will be measured by rates of successful technique among all performance. Technical success is defined as complete obliteration of the branch of splenic artery and absence of Doppler flow on EUS, and functional success, defined as improved hematologic parameters and the detectable splenic infarction by CT.

CONTACTS AND LOCATIONS:
Overall Officials: Qian Chen, Ph.D, M.D, Principal Investigator — Tongji Hospital; Zhen-gang Zhang, Ph.D, M.D, Study Chair — Tongji Hospital; Bin Cheng, Ph.D, M.D, Study Chair — Tongji Hospital
Locations (1):
- The Division of Gastroenterology, Department of Internal Medicine at Tongji Hospital, , Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei, China